CLINICAL TRIAL: NCT01449565
Title: Extended-Release Naltrexone (XR-NTX, VIVITROL) for the Treatment of Actively-Using Methamphetamine-Dependent Men Who Have Sex With Men
Brief Title: Extended-Release Naltrexone to Treat Methamphetamine Dependence in Men Who Have Sex With Men (MSM)
Acronym: TREX
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: San Francisco Department of Public Health (Other Government)
Collaborators: Alkermes, Inc. (Industry); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Phillip Coffin, MD, MIA, Director, Substance Use Research Unit, San Francisco Department of Public Health
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: R01DA031678 (NIH); R01DA031678 (NIH)
Record Dates: First submitted 2011-10-04; First posted 2011-10-10 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Amphetamine-Related Disorders
Keywords: methamphetamine; high-risk sexual behavior; HIV prevention
MeSH Terms: conditions — Amphetamine-Related Disorders | interventions — Naltrexone; vivitrol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Naltrexone (Active Comparator)
  Interventions: Drug: Naltrexone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Naltrexone — 3 monthly intramuscular injections of naltrexone 380 mg (extended release)
  Other Names: XR-NTX; VIVITROL
  Arms: Naltrexone
Drug: Placebo — 3 monthly intramuscular injections of placebo, matched to naltrexone 380 mg (extended release)
  Arms: Placebo

SUMMARY:
Extended-release naltrexone (XR-NTX, VIVITROL) is an FDA-approved medication with efficacy in treating alcohol dependence and prevention of relapse to opioid dependence. It has shown promise in reducing relapse to amphetamine use among amphetamine-dependent, yet currently amphetamine-abstinent heterosexuals. The investigators will expand upon this promising work to determine whether monthly intramuscular injections of naltrexone will reduce methamphetamine (meth) use among actively using, meth-dependent men who have sex with men (MSM) in this double-blind randomized controlled trial of extended-release naltrexone versus placebo. The investigators will focus on MSM because of the disproportionate and intertwining epidemics of meth use and HIV in this population.

DETAILED DESCRIPTION:
The investigators will enroll 100 sexually active, meth-dependent MSM who will be randomized 1:1 to receive monthly injections of extended-release naltrexone (n=50) or placebo (n=50) for 12 weeks at weeks 0, 4, and 8. Study participants will be seen weekly at our site at the HIV Prevention Section of the San Francisco Department of Public Health, where they will provide urine for drug testing and participate in substance use counseling. All participants will receive HIV risk-reduction counseling. Behavior will be assessed using standardized measures via audio computer-assisted self-interview (ACASI).

ELIGIBILITY:
Inclusion criteria:

1. born male; or born female and does not identify as female
2. reports having anal sex with men in the prior six months while under the influence of meth;
3. diagnosed with meth dependence as determined by SCID;
4. interested in stopping or reducing meth use;
5. at least one meth-positive urine during screening and run-in period;
6. no current acute illnesses requiring prolonged medical care;
7. no chronic illnesses that are likely to progress clinically during trial participation;
8. able and willing to provide informed consent and adhere to visit schedule;
9. age 18-65 years;
10. baseline CBC, total protein, albumin, glucose, alkaline phosphatase, creatinine, BUN, total bilirubin, and electrolytes without clinically significant abnormalities as determined by investigator in conjunction with symptoms, physical exam, and medical history.

Exclusion criteria:

1. any psychiatric condition (e.g. current depression with suicidal ideation or schizophrenia) that would preclude safe participation in the protocol;
2. known intolerance and/or hypersensitivity to naltrexone, carboxymethylcellulose, or polylactide-co-polymers (PLG) or any other components of the diluents;
3. current use of or dependence on any opioids; a known medical condition which currently requires or is likely to require opioid analgesics; or positive opioid urine screening tests
4. diagnosed with current alcohol dependence as determined by the SCID;
5. current CD4 count < 200 cells/mm3;
6. moderate or severe liver disease (AST and/or ALT > 5 times upper limit of normal);
7. moderately or severely impaired renal function (eGFR < 50 mL/min);
8. thrombocytopenia or other coagulation disorder
9. currently participating in another research study;
10. pending legal proceedings with high risk for incarceration during the time of planned study participation;
11. any condition that, in the principal investigator's judgment, interferes with safe study participation or adherence to study procedures.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2012-09; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
urine meth positivity | 12 weeks
  proportion of meth-metabolite positive urines by study arm, measured weekly from week 0 through week 12

SECONDARY OUTCOMES:
reduction in sexual risk behavior | 12 weeks
  reduction in meth-associated sexual risk behavior as measured by: numbers of male anal sex partners, serodiscordant condomless anal sex partners, serodiscordant condomless anal sex events, serodiscordant condomless receptive anal sex partners, serodiscordant condomless receptive anal sex events, serodiscordant condomless insertive anal sex partners, serodiscordant condomless insertive anal sex events, and numbers of sex partners with whom meth was used, by study arm
percentage of total expected injections administered | 12 weeks
  acceptability of extended-release naltrexone vs placebo, as measured by the percentage of total expected injections administered, by study arm
rates of adverse events | 12 weeks
  rates of adverse events will be compared by study arm

CONTACTS AND LOCATIONS:
Overall Officials: Steven L. Batki, MD, Principal Investigator — Substance Abuse Programs, San Francisco VA Medical Center; Phillip Coffin, MD, MIA, Principal Investigator — Substance Use Research Unit, San Francisco Department of Public Health; Emily Behar, MS, Study Director — San Francisco Department of Public Health
Locations (1):
- Substance Use Research Unit, San Francisco, California, United States